CLINICAL TRIAL: NCT04333225
Title: A Prospective Clinical Study of Hydroxychloroquine in the Prevention of SARS- CoV-2 (COVID-19) Infection in Healthcare Workers After High-risk Exposures
Brief Title: Hydroxychloroquine in the Prevention of COVID-19 Infection in Healthcare Workers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 020-132
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Results first posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: hydroxychloroquine
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine (Experimental): Subjects who chose to enter the HCQ arm received a loading dose of 800 mg HCQ on day 1 followed by two 200 mg tablets once a week for a total of 7 weeks
  Interventions: Drug: Hydroxychloroquine
- Control (No Intervention): Subjects who declined taking HCQ were considered as controls

INTERVENTIONS:
Drug: Hydroxychloroquine — Weekly treatment in individuals at high risk
  Other Names: Plaquenil; HCQ
  Arms: Hydroxychloroquine

SUMMARY:
In order to assess the efficacy of hydroxychloroquine treatment weekly for a total of 7 weeks in the prevention of COVID-19 infection, three hundred sixty (360) Healthcare workers with high risk exposure to patients infected with COVID-19 will be tested for COVID-19 infection via nasopharyngeal (NP) swab once weekly for 7 weeks. Of those, one hundred eighty (180) will receive weekly doses of hydroxychloroquine for the duration of the study. Subjects who opt not to receive the study drug will form the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and female healthcare workers ≥ 18 to ≤ 75 years of age upon study consent
2. Healthcare workers with

   • One day or more of exposure to suspect and/or positive COVID-19 patients, including but not limited to those working in the Emergency Department or Intensive Care Unit.

   OR

   • Unprotected exposure to a known positive COVID-19 patient within 72 hours of screening.
3. Afebrile with no constitutional symptoms
4. Willing and able to comply with scheduled visits, treatment plan, and other study procedures
5. Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study prior to initiation of any subject-mandated procedures

Exclusion Criteria:

1. Participation in other investigational clinical trials for the treatment or prevention of SARS-COV-2 infection within 30days
2. Unwilling to practice acceptable methods of birth control (both males who have partners of childbearing potential and females of childbearing potential) during Screening, while taking study drug, and for at least 30 days after the last dose of study drug is ingested Note: the following criteria follow standard clinical practice for FDA approved indications of this medication
3. Having a prior history of blood disorders such as aplastic anemia, agranulocytosis, leukopenia, or thrombocytopenia
4. Having a prior history of glucose-6-phosphate dehydrogenase (G-6-PD) deficiency
5. Having dermatitis, psoriasis or porphyria
6. Taking Digoxin, Mefloquine, methotrexate, cyclosporine, praziquantel, antacids and kaolin, cimetidine, ampicillin, Insulin or antidiabetic drugs, arrhythmogenic drugs, antiepileptic drugs, loop, thiazide, and related diuretics, laxatives and enemas, amphotericin B, high dose corticosteroids, and proton pump inhibitors, neostigmine, praziquantel, Pyridostigmine, tamoxifen citrate
7. Allergies: 4-Aminoquinolines
8. Pre-existing retinopathy of the eye
9. Has a chronic liver disease or cirrhosis, including hepatitis B and/or untreated hepatitis
10. Untreated or uncontrolled active bacterial, fungal infection
11. Known or suspected active drug or alcohol abuse, per investigator judgment
12. Women who are pregnant or breastfeeding
13. Known hypersensitivity to any component of the study drug
14. A known history of prolonged QT syndrome or history of additional risk factors for torsades de pointe (e.g., heart failure, requires a lab test , family history of Long QT Syndrome), or the use of concomitant medications that prolong the QT/QTc interval

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A McCullough, MD, MPH, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All study subjects were employed by and worked at the Baylor University Medical Center in Dallas, Texas.
Period: Overall Study
Arm/Group | Hydroxychloroquine | Control
Started | 101 | 120
Completed | 98 | 115
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydroxychloroquine | Control | Total
Number analyzed (Participants) | 101 | 120 | 221
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.90 (12.42) | 34.53 (800) | 35.36 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 101 | 167
  Male | 35 | 19 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 26 | 42
  Not Hispanic or Latino | 85 | 94 | 179
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 4 | 4 | 8
  White | 78 | 104 | 182
  Others | 19 | 12 | 31
Region of Enrollment [Number; unit: participants]
  United States | 101 | 120 | 221
Cough score [Mean (Standard Deviation); unit: Millimeters] — Cough Visual Analogue Scale was recorded at baseline to assess cough severity in patients. Each patient was asked to mark on a 100 mm scale between 0 representing 'no cough' and 100 representing the 'worst cough'.
  Millimeters | 2.74 (7.66) | 3.26 (7.46) | 3.02 (7.54)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Infected With COVID-19 or COVID-19 Like Illness During the Trial
Description: Number of participants infected with COVID-19 or identified as having COVID-19 like illness during the trial
Time Frame: Up to 7 weeks after study initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Control
Number analyzed (Participants) | 101 | 120
Participants | 13 | 32
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Control; Test type: Other — Other: estimating risk reduction; p = 0.0112, Chi-squared; Risk Ratio (RR) = 2.0718, 95% CI 2-sided [1.15 to 3.72]

2. Secondary Outcome: Time From Study Initiation Until the Occurrence of COVID-19 or COVID-19 Like Illness or Being Censored
Description: Time-to-first clinical event consisting of a persistent change for any of the following:
  * diagnosis of COVID-19
  * clinical characteristics of COVID-19 like illness
  * being censored
Time Frame: Up to 7 weeks after study initiation
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Hydroxychloroquine | Control
Number analyzed (Participants) | 101 | 120
Days | 43.17 (11.15) | 39.25 (15.02)
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Control; Test type: Other — Other: Estimating hazard ratio; p = 0.0105, Log Rank; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.17 to 0.75]

ADVERSE EVENTS:
Time Frame: 7 weeks
Arm/Group | Hydroxychloroquine | Control
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/120
Serious Adverse Events (participants affected / at risk) | 1/101 | 0/120
Other Adverse Events (participants affected / at risk) | 21/101 | 0/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine (N=101) | Control (N=120)
COVID-19 like illness (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine (N=101) | Control (N=120)
Nausea (Gastrointestinal disorders) | 13 (21) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 8 (21) | 0 (0)

LIMITATIONS AND CAVEATS:
* Due to the off-label use of HCQ, we were not able to incorporate randomization in our design.
* The outcome of CLI was based on self-reported symptoms, which is prone to bias.
* The trial may be under-powered as recruitment was forced to stop early at 221 instead of 360 because of the demand for and subsequent shortage of HCQ in March 2020.
* Our study participants were young and healthy compared to other prophylaxis trials, which may partially explain the low rates of COVID-19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/25/NCT04333225/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/25/NCT04333225/SAP_001.pdf